CLINICAL TRIAL: NCT04133753
Title: Evaluating Effectiveness of a Communication Facilitator to Reduce Distress and Improve Goal Concordant Care for Critically Ill Patients and Their Families: A Randomized Trial. Famiréa - FCS
Brief Title: Evaluating Effectiveness of a Communication Facilitator : A Randomized Trial
Acronym: Famirea - FCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: APHP180586
Record Dates: First submitted 2019-10-18; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Intensive Care Unit; Life Stress; Family Members; Facilitation, Social
MeSH Terms: conditions — Stress, Psychological; Social Facilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facilitator-Based Intervention (Experimental): The 'Facilitator-Based Intervention' includes patient and family member subjects.
  Interventions: Behavioral: Facilitator-Based Intervention
- Usual Care (No Intervention): The 'Usual Care' arm includes patient and family member subjects.

INTERVENTIONS:
Behavioral: Facilitator-Based Intervention — Facilitators interact in person with patients, family, and clinicians both during and following the patient's ICU stay for 3 months. In-person contacts include visits to patients' homes and/or care facilities; phone contacts include calls to patients, families and clinicians. Patients and families have access to facilitators through phone and email. Facilitators may attend clinic visits with patients. In addition to checking directly with patients/families during regular contacts, facilitators also access the electronic health record to ensure they have accurate information about appointments and treatment plans and to document key points for the clinical team. Facilitators encourage referral to inpatient or outpatient palliative care services when needs are identified.
  Other Names: Communication Facilitator
  Arms: Facilitator-Based Intervention

SUMMARY:
This study is a randomized clinical trial of an intervention to improve outcomes for patients and their family by using ICU nurse facilitators to support, model, and teach communication strategies that enable patients and their families to secure care in line with patients' goals of care over an illness trajectory, beginning in the ICU and continuing to care in the community.

DETAILED DESCRIPTION:
The impact of critical illness is increasing due to an aging population as well as advances in effectiveness and availability of critical care. Critically ill patients and their families suffer a high burden of symptoms of depression, anxiety, and post-traumatic stress due, in part, to fragmented medical care that is often poorly aligned with their goals. Fragmented care includes numerous transitions for patients and families across clinicians and across settings, starting in the intensive care unit (ICU) and extending to acute care, skilled nursing facilities, or home. As illness progresses, patients and families struggle to navigate the spectrum of goals of care, to match their values and goals with treatments, to communicate their goals to their clinicians, and to make difficult medical decisions without letting unmet emotional needs interfere. Poor communication exacerbated by these transitions compounds an already stressful experience, causing distress to patients and their families. Taken together, these issues lead to ineffective communication during and after the ICU which can often result in high intensity "default" care that may be unwanted.

Using a randomized trial, this project aims to evaluate an innovative model of care in which ICU nurse facilitators support, model, and teach communication strategies that enable patients and families to secure care in line with their goals over an illness trajectory, beginning in the ICU and continuing into the community. Facilitators use communication skills, attachment theory, and mediation to improve: 1) patients' and families' self-efficacy to communicate with clinicians within and across settings; 2) patients' and families' outcome expectation that communication with clinicians can improve their care; and 3) patients' and families' behavioral capability through skill building to resolve barriers to effective communication and mediate conflict. Facilitators work with seriously ill patients and their families beginning with a critical care unit stay and following them over the course of three months.

The intervention's effectiveness will be measured with patient- and family-centered outcomes at 1-, 3-, and 6-months post-randomization. The primary outcome is family members' burden of symptoms of depression over the 6 months. The investigators also evaluate whether the intervention improves the value of healthcare by reducing healthcare costs while improving patient and family outcomes. Finally, investigators use qualitative methods to explore implementation factors (intervention, settings, individuals, processes) associated with improved implementation outcomes (acceptability, fidelity, penetration) to inform dissemination of this type of intervention to support patients and their families. This study aims to address key knowledge gaps while evaluating a methodologically rigorous intervention to improve outcomes for patients with serious illness and their families across the trajectory of care and the spectrum of goals of care.

ELIGIBILITY:
Inclusion Criteria:

Patient:

* Age >=18 years
* Admitted to the ICU with an expected length of stay of at least 2 days
* A chronic life-limiting illness suggesting a median survival of approximately 2 years or a risk of hospital mortality of >15% using either SOFA score, APACHE score or Injury Severity Score (with any one or more score predicting hospital mortality >15%)
* Patient informed consent or relative or trusted person of patient consent (when lacking patient decisional capacity)
* Patient with visiting relatives

Family member:

* Age >=18 years
* Family will be identified by the patient. If the patient does not have decisional capacity, family will be identified by a legal surrogate decision-maker. We will not limit the number of family members who can participate but anticipate 1-3 family members per patient (average 1.5 based on prior studies).
* Family informed consent

Exclusion Criteria:

Patient:

* Non-French speaking patient or relative
* Pregnant or breastfeeding patient
* No social security coverage Family Member
* Non-French speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) - family | 6 months after randomization
  Family member symptoms of depression and anxiety assessed with the Hospital Anxiety and Depression Scale (HADS), which has become standard for ICU and post-ICU studies. The HADS is a reliable and valid 14-item, 2-domain (anxiety and depression) tool used to assess symptoms of psychological distress. Seven items evaluate anxiety and seven evaluate depression. Each item is scored on a 4-point scale (ranging from 0-3) with scores for each subscale (anxiety and depression) ranging from 0-21. HADS has been used in over 700 studies with evidence of reliability, validity and responsiveness among critically ill patients and their family.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) - family 1, 3 | 1- and 3- months after randomization
  Family member symptoms of depression and anxiety assessed with the Hospital Anxiety and Depression Scale (HADS), which has become standard for ICU and post-ICU studies. The HADS is a reliable and valid 14-item, 2-domain (anxiety and depression) tool used to assess symptoms of psychological distress. Seven items evaluate anxiety.
Hospital Anxiety and Depression Scale (HADS) - patient 1, 3, 6 | 1-, 3-, and 6-months after randomization
  Patient symptoms of depression and anxiety assessed with the Hospital Anxiety and Depression Scale (HADS), which has become standard for ICU and post-ICU studies. The HADS is a reliable and valid 14-item, 2-domain (anxiety and depression) tool used to assess symptoms of psychological distress. Seven items evaluate anxiety and seven evaluate depression. Each item is scored on a 4-point scale (ranging from 0-3) with scores for each subscale (anxiety and depression) ranging from 0-21. HADS has been used in over 700 studies with evidence of reliability, validity and responsiveness among critically ill patients and their family.
Hospital Anxiety and Depression Scale - Anxiety subscale - family 1, 3, 6 | 1-, 3-, and 6-months after randomization
  Family member symptoms of depression and anxiety assessed with the Hospital Anxiety and Depression Scale (HADS), which has become standard for ICU and post-ICU studies. The HADS is a reliable and valid 14-item, 2-domain (anxiety and depression) tool used to assess symptoms of psychological distress. Seven items evaluate anxiety.
Hospital Anxiety and Depression Scale - Anxiety subscale - patient 1, 3, 6 | 1-, 3-, and 6-months after randomization
  Patient symptoms of depression and anxiety assessed with the Hospital Anxiety and Depression Scale (HADS), which has become standard for ICU and post-ICU studies. The HADS is a reliable and valid 14-item, 2-domain (anxiety and depression) tool used to assess symptoms of psychological distress. Seven items evaluate anxiety.
Goal-concordant care (SUPPORT items) - patient and family | 1-, 3-, and 6-months after randomization
  Concordance between the care patients want and the care they are receiving will be measured with two questions from the SUPPORT study. The first defines patients' preferences: "If the patient had to make a choice at this time, would the patient prefer a course of treatment focused on extending life as much as possible, even if it means having more pain and discomfort, or would the patient want a plan of care focused on relieving pain and discomfort as much as possible, even if that means not living as long?" The second question assesses perceptions of current treatment using the same two options. The outcome is a dichotomous variable of whether the preference matches the report of care received. Although this creates a "false dichotomy" in that many patients want both, this "forced choice" helps identify patients' top priority. Based on prior studies, we expect only 50-60% of controls will report goal-concordant care.
PTSD Checklist-Civilian (PCL) - Post-traumatic Stress Symptoms - patient | 1-, 3-, and 6-months after randomization
  The PTSD Checklist-Civilian (PCL) uses 17 self-report items to assess the intrusive, avoidant, and arousal PTSD symptom clusters. Responses are recorded on a 5 points scale that ranges from "not at all" to "extremely". The measure can be scored continuously or for symptoms consistent with a diagnosis of PTSD. The measure is reliable and valid across diverse populations. It has also demonstrated responsiveness in a randomized trial of stepped collaborative care for trauma survivors.
PTSD Checklist-Civilian (PCL) - Post-traumatic Stress Symptoms - family | 1-, 3-, and 6-months after randomization
  The PTSD Checklist-Civilian (PCL) uses 17 self-report items to assess the intrusive, avoidant, and arousal PTSD symptom clusters. Responses are recorded on a 5 points scale that ranges from "not at all" to "extremely". The measure can be scored continuously or for symptoms consistent with a diagnosis of PTSD. The measure is reliable and valid across diverse populations. It has also demonstrated responsiveness in a randomized trial of stepped collaborative care for trauma survivors.
QUAL-E - patient | 1-, 3-, and 6-months after randomization
  Measuring the quality of life of seriously ill patients. The QUAL-E is a validated instrument with ~25 items measuring of quality of life at the end of life with a four-domain structure: life completion, symptoms impact, relationship with health care provider, and preparation for end of life.
QUAL-E - family | 1-, 3-, and 6-months after randomization
  Measure of family experience of patients with serious illness. The QUAL-E (Fam) is a validated ~17-item companion instrument to the patient QUAL-E measure of quality of life at the end of life.
Perceived Health Competence Scale (PHCS) - family | 1-, 3-, and 6-months after randomization
  We will use the Perceived Health Competence Scale (PHCS), an 8-item questionnaire assesses family self-efficacy, outcome expectations, and behavioral capacity for healthcare. It has been used to predict health behaviors and outcomes in older adults, people with chronic disease, women with breast cancer, and patients in dialysis. It has internal consistency reliability from 0.82-0.90. Construct validity was supported with a single factor structure underlying the total score and concurrent validity was supported by significant correlations with health status. It is a mediator of psychosocial outcomes and found to be an important explanatory variable linking access to information and psychosocial health outcomes.
Perceived Health Competence Scale (PHCS) - patient | 1-, 3-, and 6-months after randomization
  We will use the Perceived Health Competence Scale (PHCS), an 8-item questionnaire assesses patient self-efficacy, outcome expectations, and behavioral capacity for healthcare. It has been used to predict health behaviors and outcomes in older adults, people with chronic disease, women with breast cancer, and patients in dialysis. It has internal consistency reliability from 0.82-0.90. Construct validity was supported with a single factor structure underlying the total score and concurrent validity was supported by significant correlations with health status. It is a mediator of psychosocial outcomes and found to be an important explanatory variable linking access to information and psychosocial health outcomes.
SF-1 - Health related quality of life - family | 1-, 3-, and 6-months after randomization
  We will use the SF-1 on family members, a shorter version of the functional health status scale adapted from the SF12 which has been used with patients with chronic illness and with older populations, and has good psychometric characteristics including internal reliability (Cronbach alphas >=0.70), test-retest reliability (r>0.73), and validity supported by confirmatory factor analysis and hypothesis testing.
SF-1 - Health related quality of life - patient | 1-, 3-, and 6-months after randomization
  We will use the SF-1 on patients, a shorter version of the functional health status scale adapted from the SF12 which has been used with patients with chronic illness and with older populations, and has good psychometric characteristics including internal reliability (Cronbach alphas >=0.70), test-retest reliability (r>0.73), and validity supported by confirmatory factor analysis and hypothesis testing.
ICU length of stay | 6-months after randomization
  Delay between randomization and ICU discharge
Hospital length of stay | 6-months after randomization
  Delay between randomization and hospital discharge

OTHER OUTCOMES:
Qualitative interviews | 6-months after randomization
  Qualitative interviews to evaluate components of the intervention and explore barriers and facilitators to implementation of the intervention.
return to work - family | 6-months after randomization
  delay between randomization and return to work for family members
return to work - patient | 6-months after randomization
  delay between randomization and return to work for patients
hospital utilization after hospital discharge | 6-months after randomization
  We will also estimate incidence of hospital utilization after hospital discharge in exploratory analyses, including readmissions and emergency department visits over 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Louis Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Renet A, Azoulay E, Reignier J, Cariou A, Renault A, Huet O, Pochard F, Engelberg RA, Kentish-Barnes N. "It's all about setting the stage." The nurse facilitator trial: perceived outcomes and implementation issues. A qualitative study among ICU clinicians and nurse facilitators. Intensive Care Med. 2024 Oct;50(10):1657-1667. doi: 10.1007/s00134-024-07589-z. Epub 2024 Aug 19. PMID 39158706
- [Derived] Kentish-Barnes N, Azoulay E, Reignier J, Cariou A, Lafarge A, Huet O, Gargadennec T, Renault A, Souppart V, Clavier P, Dilosquer F, Leroux L, Lege S, Renet A, Brumback LC, Engelberg RA, Pochard F, Resche-Rigon M, Curtis JR. A randomised controlled trial of a nurse facilitator to promote communication for family members of critically ill patients. Intensive Care Med. 2024 May;50(5):712-724. doi: 10.1007/s00134-024-07390-y. Epub 2024 Apr 4. PMID 38573403